CLINICAL TRIAL: NCT03341299
Title: A Study to Evaluate the Pharmacokinetics and Glucodynamics of LY900014 Compared to Humalog® in Patients With T1DM
Brief Title: A Comparative Study of LY900014 With Insulin Lispro (Humalog) in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16641; I8B-MC-ITRV (Other: Eli Lilly and Company); 2017-001500-30 (EudraCT Number)
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LY900014 Before Meal (Experimental): Individualized dose of LY900014 administered subcutaneously (SC) immediately before meal in one of four study periods.
  Interventions: Biological: LY900014
- LY900014 After Meal (Experimental): Individualized dose of LY900014 administered SC 20 minutes after start of meal in one of four study periods.
  Interventions: Biological: LY900014
- Insulin Lispro (Humalog) Before Meal (Active Comparator): Individualized dose of insulin lispro administered SC immediately before meal in one of four study periods.
  Interventions: Biological: Insulin Lispro
- Insulin Lispro (Humalog) After Meal (Active Comparator): Individualized dose of insulin lispro administered SC 20 minutes after start of meal in one of four study periods.
  Interventions: Biological: Insulin Lispro

INTERVENTIONS:
Biological: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 After Meal; LY900014 Before Meal
Biological: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog) After Meal; Insulin Lispro (Humalog) Before Meal

SUMMARY:
The purpose of this study is to evaluate a new formulation of insulin lispro, LY900014, which is a drug that lowers blood sugar. The study will look at how the body processes LY900014, and the effect of LY900014 on blood sugar levels following a standard meal. For each participant, the study will consist of 4 periods and there will be approximately 12 weeks from screening to final study follow up.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with Type 1 Diabetes Mellitus (T1DM) for at least 1 year
* Have a body mass index (BMI) of 18.5 kilogram per meter square (kg/m²) to 35.0 kg/m²
* Have a glycated hemoglobin (HbA1c) ≤9.0% at screening
* Are on stable prandial insulin and basal insulin (neutral protamine Hagedorn [NPH] insulin, insulin glargine or insulin detemir) for at least 3 months before screening with a total insulin dose demand of less than or equal to (≤) 1.5 units per kilogram per day (U/kg/day)

Exclusion Criteria:

* Are currently enrolled, or have participated within the last 30 days, in a clinical trial or any other type of medical research
* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate in the study
* Have donated blood of more than 450 millilitre (mL) or more in the last 3 months or provided any blood donation within the last month before screening.
* Any significant changes in insulin regimen and/or unstable blood glucose control within the past 3 months prior to screening as assessed by the investigator.
* Are treated with a CSII (insulin pump)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Individualized dose of LY900014 or insulin lispro (Humalog) administered subcutaneously (SC) with 21 hours between doses
  Period 1: LY900014 administered subcutaneously (SC) immediately before meal Period 2: insulin lispro (Humalog) administered SC 20 minutes after start of meal Period 3:LY900014 administered SC 20 minutes after start of meal Period 4: insulin lispro administered SC immediately before meal
- Cohort 2: Individualized dose of LY900014 or insulin lispro (Humalog) administered subcutaneously (SC) with 21 hours between doses
  Period 1:LY900014 administered SC 20 minutes after start of meal Period 2: LY900014 administered subcutaneously (SC) immediately before meal Period 3: insulin lispro (Humalog) administered SC immediately before meal Period 4: insulin lispro (Humalog) administered SC 20 minutes after start of meal
- Cohort 3: Individualized dose of LY900014 or insulin lispro (Humalog) administered subcutaneously (SC) with 21 hours between doses
  Period 1: insulin lispro (Humalog) administered SC immediately before meal Period 2:LY900014 administered SC 20 minutes after start of meal Period 3: insulin lispro (Humalog) administered SC 20 minutes after start of meal Period 4: LY900014 administered subcutaneously (SC) immediately before meal
- Cohort 4: Individualized dose of LY900014 or insulin lispro (Humalog) administered subcutaneously (SC) with 21 hours between doses
  Period 1: insulin lispro (Humalog) administered SC 20 minutes after start of meal Period 2: insulin lispro (Humalog) administered SC immediately before meal Period 3: LY900014 administered subcutaneously (SC) immediately before meal Period 4:LY900014 administered SC 20 minutes after start of meal
Period: Period 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout (A Minimum of 21 Hours)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout (A Minimum of 21 Hours)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout (A Minimum of 21 Hours)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Overall Study: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 36
Duration of Type 1 Diabetes Mellitis [Mean (Standard Deviation); unit: years] | 21.41 (13.60)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve (AUC)
Description: PK: Insulin Lispro AUC for Each Treatment Arm. LY900014 before and after meal and insulin lispro (Humalog) before and after meal were pooled by treatment to evaluate the overall PK of LY900014 and insulin lispro (Humalog) per protocol .
Time Frame: Predose, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, and 420 minutes (7 hours)
Population: All randomized participants who received at least 1 dose of study drug. LY900014 before and after meal and insulin lispro (Humalog) before and after meal were pooled by treatment to evaluate the overall PK of LY900014 and insulin lispro (Humalog) per protocol .
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles times hour per Liter
Groups:
- LY900014: All participants who received individualized dose of LY900014 SC before meal or 20 minutes after start of meal
- Insulin Lispro (Humalog): All participants who received individualized dose of insulin lispro (Humalog) SC before meal or 20 minutes after start of meal
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 35 | 35
picomoles times hour per Liter | 970 (57) | 968 (56)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.7734, Mixed Models Analysis; Ratio of geometric least square means = 0.991, 95% CI 2-sided [0.932 to 1.05]

2. Secondary Outcome: Glucodynamics (GD): Area Under the Baseline Subtracted Glucose Concentration Curve
Description: GD: Area Under The Baseline Subtracted Glucose Concentration Curve for Each Treatment Arm
Time Frame: Predose, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, and 300 minutes postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable glucodynamic parameters.
Measure: Mean (Standard Deviation); unit: milligrams times hour per deciLiter
Groups:
- Insulin Lispro (Humalog) Before Meal: Individualized dose of insulin lispro (Humalog) administered SC immediately before meal in one of four study periods.
Arm/Group | LY900014 Before Meal | LY900014 After Meal | Insulin Lispro (Humalog) Before Meal | Insulin Lispro (Humalog) After Meal
Number analyzed (Participants) | 30 | 29 | 32 | 29
milligrams times hour per deciLiter | 207 (189) | 264 (205) | 227 (163) | 327 (212)
Statistical Analysis 1: Comparison: LY900014 Before Meal vs Insulin Lispro (Humalog) Before Meal; Test type: Superiority; p = 0.7190, Mixed Models Analysis; difference in LS means = -14.50, 95% CI 2-sided [-94.38 to 65.38]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: All participants who received at least 1 dose of study drug.
Groups:
- Insulin Lispro (Humalog) After Meal: Individualized dose of insulin lispro (Humalog) administered SC 20 minutes after start of meal in one of four study periods.
Arm/Group | LY900014 Before Meal | LY900014 After Meal | Insulin Lispro (Humalog) Before Meal | Insulin Lispro (Humalog) After Meal
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 3/35 | 3/36 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 Before Meal (N=35) | LY900014 After Meal (N=35) | Insulin Lispro (Humalog) Before Meal (N=36) | Insulin Lispro (Humalog) After Meal (N=35)
Injection Site Reaction (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03341299/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03341299/SAP_001.pdf